## MODULATION OF AIRWAY REACTIVITY WITH CHRONIC MECHANICAL STRAIN

# **Principal Investigator:**

Robert S. Tepper, MD, PhD

705 Riley Hospital Drive, ROC 4270 Indianapolis, IN 46202

# **Co-Investigators:**

Susan Gunst, Ph.D. Hasna Jalou, M.D. Nadia Krupp, M.D.

Dated: March 17, 2016

Indiana University School of Medicine

Department of Pediatrics

Pulmonology, Allergy, and Sleep Medicine

Riley Hospital for Children at Indiana University Health

# **Table of Contents:**

| <b>0</b> 4- | | O - I | nema |
|-------------|-----|-------|---------------------|
| ►TI | INV | > Cr | 10M2 |
| ULL | uuv | UUI | ı <del>c</del> ıııa |

- 1.0 Background, Rationale, and Specific Aims
- 2.0 Inclusion/Exclusion Criteria
- 3.0 Enrollment/Randomization
- 4.0 Study Procedures
- 5.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 6.0 Study Withdrawal/Discontinuation
- 7.0 Statistical Considerations
- 8.0 Privacy and Confidentiality Issues
- 9.0 Follow up and Record Retention
- 10.0 Administrative, Ethical, Regulatory Considerations

# 1.0 Background

Asthma is characterized by chronic airway inflammation, repeated episodes of reversible airway obstruction and airway hyper-reactivity. Airway inflammation and clinical symptoms of asthma are most often initiated by IgE-mediated responses following exposure to environmental allergens. Inflammatory cell recruitment into the lungs and airway hyper responsiveness are key components of the allergen-induced inflammatory response, which results from the interaction of resident airway cells and inflammatory cells that release local mediators. Patients with severe, recurrent asthma also have remodeling of the airway wall with increased airway smooth muscle, increased inflammatory cells and collagen deposition.

For many decades, corticosteroids have been used to control airway inflammation, while  $\beta$ -adrenergic bronchodilators have been the primary treatment for bronchoconstriction. Although these therapies are effective for the vast majority of asthmatics, they are limited by high cost, poor adherence, and increasing concern about long-term adverse effects. The FDA has issued a black-box warning linking long-acting  $\beta$ - adrenergic bronchodilators to asthma deaths, and other studies have linked corticosteriods to fracture risk and growth retardation 10-12. Recently introduced therapies that focus on inhibiting a single component of the allergic inflammatory response, such as anti-IL-5 or anti-IL-13 antibodies, have had limited efficacy 13. Thus, there is a compelling need for new, safe and effective approaches to asthma treatment, particularly in children with severe asthma, where there is generally a lifelong burden of disease, use of medications, and accounts for the majority of health care expenditures among all children with asthma. The development of a therapeutic approach that could reduce both airway responsiveness and airway inflammation would be an important advance in the treatment of asthma.

During the previous funding period of this project, our laboratory demonstrated that chronic mechanical strain imposed on the airways *in vivo* using continuous positive airway pressure (CPAP) results in a dramatic reduction in airway reactivity *in vivo* in mice, ferrets and rabbits<sup>1-3</sup>. Lungs, airways and airway smooth muscle (ASM) tissues isolated from CPAP-treated animals studied *in vitro* exhibited lower responsiveness to bronchoconstrictors<sup>1-3</sup>. We also observed this suppression of airway responsiveness by chronic mechanical strain in a rabbit model of allergic asthma<sup>5</sup>. These animal studies led to a small clinical trial in which adults with asthma were treated with nocturnal CPAP for 1 week. CPAP caused a significant reduction in airway reactivity in these patients<sup>6</sup>. This novel approach for treating airway hyper-reactivity is currently being evaluated in a NIH multi-center Phase II clinical trial of adults with mild to moderate asthma (U01 HL108730).

We now propose to determine the efficacy of chronic mechanical strain as an inhibitor of airway inflammation. Our preliminary studies have demonstrated that chronic mechanical strain can suppress the responses of airway tissues to allergic inflammatory stimuli and suppress the activation of signaling molecules involved in these responses<sup>3,14,15</sup>. Based on these studies, we hypothesize that chronic mechanical strain will inhibit signaling processes in airway tissues that lead to airway inflammation, hyper-reactivity and remodeling. We propose a novel molecular mechanism for the inhibitory effects of chronic mechanical strain on the responses of ASM to inflammatory stimuli. Anti-inflammatory agents such as corticosteroids remain the primary treatment for severe chronic asthma. The consequences of long term steroid therapy can be extremely deleterious, particularly in children, for whom steroids can have a significant adverse impact on growth and development. Our proposed study will provide the basis for a new non-pharmacologic therapy for the control of asthma that may be particularly important for the treatment of children with severe steroid-dependent disease. We will determine whether mechanical strain, as delivered using CPAP, is an effective therapy for suppressing airway hyper-reactivity and inflammation in pediatric subjects with severe asthma. The concept that a non-pharmacologic therapy may play such a pivotal role in suppressing ASM contraction, inflammation and tissue remodeling is novel and exciting. Furthermore, elucidation of the molecular mechanisms by which strain suppresses inflammatory signaling pathways could also provide a basis for the development of new pharmacologic targets for asthma therapy.

**Pathophysiology of airway inflammation in asthma.** Th2 cytokines derived from CD4+ T lymphocytes play a pivotal role in the airway pathology associated with asthma<sup>16-19</sup>. The structurally related Th2 cell derived cytokines interleukin (IL)-4 and IL-13 stimulate allergic and eosinophilic inflammation as well as

epithelial and smooth muscle changes, and they are widely recognized as mediators of allergen-induced airway hyperresponsiveness and airway remodeling<sup>8,18-21</sup>. Th2 cytokines can induce airway hyperreactivity without inflammatory cell recruitment which indicates that many of the pathophysiologic effects of allergic inflammation in asthma result from the direct actions of IL-4 or IL-13 on airway cells<sup>9,19,20,22-24</sup>. The incubation of ASM with IL-

13 or IL-4 *in vitro* causes ASM hypercontractility, inhibits relaxation to isoproterenol and stimulates release of the eosinophil chemo-attractant eotaxin and IL-5<sup>7,9,25-28</sup>. The cytokines secreted by ASM and other airway cells have paracrine effects on inflammatory cells and thus contribute to airway inflammation<sup>29-31</sup>.

Phenotypic alterations in airway cells induced by the direct actions of cytokines may be a primary mechanism for airway remodeling in asthma. Changes in gene expression induced by IL-13 or IL-4 have been demonstrated in airway cells including ASM, fibroblasts and airway epithelial cells<sup>15,32,33</sup>. Both IL-4 and IL-13 activate signaling pathways that regulate cell growth and proliferation as well as the expression of responsive genes<sup>34</sup>. The direct stimulation of resident airway cells with inflammatory cytokines *in vitro* stimulates cell growth and proliferation and the secretion of matrix proteins<sup>13,35,36</sup>. *In our previous animal studies, , we evaluated the effects of chronic mechanical strain on the physiologic responses of ASM tissues to inflammatory mediators in vitro, and on airway inflammation and remodeling in vivo using murine models of asthma.* 

#### Molecular mechanisms for the direct effects of inflammatory cytokines on ASM cells.

IL-4 and IL-13 both signal through a heterodimeric receptor complex that consists of an IL-4Rα chain and an IL-13Rα chain (Fig.1). In response to stimulation, the IL-4/IL-13 receptor subunits associate with Janus kinases (Jak) that phosphorylate the IL4Rα and IL13 receptor side chains, activating two distinct signaling proteins that bind to the phosphorylated IL-4Rα receptor side chain: insulin receptor-2 (IRS-2) and "signal transducer and activator of transcription 6"(STAT6)34. IRS2 activates the PI3 kinase-dependent protein kinase Akt, a regulator of cell growth and hypertrophy, as well as ERK1/2 MAP kinase and other MAP kinases. phosphorylation by Jak, activated STAT6 dimerizes and migrates to the nucleus where it initiates the transcription of IL-4/IL-13 responsive genes. Stimulation of ASM cells or tissues by IL-4/IL-13 in vitro results in the phosphorylation of Akt, ERK1/2 and STAT6, the and synthesis



secretion of eotaxin and IL-5, and suppresses the expression of smooth muscle phenotype-specific proteins<sup>7,8,15,26,37-40</sup> (Figs.1,4-6). Our previous studies and preliminary data have shown that chronic mechanical strain suppresses the activation of Akt and ERK, and that strain inhibits eotaxin secretion and IL-13-mediated gene transcription (Figs. 5,6,9).

#### Chronic mechanical strain suppresses airway responsiveness and ASM contractility.

Mechanical strain of the lungs during breathing has an important role in reducing airway responsiveness<sup>41</sup>. Deep inspirations and tidal breathing decrease airway responsiveness acutely in healthy adults and animals and their absence increases airway responsiveness<sup>42-47</sup>. Similar effects of mechanical strain have been observed in isolated airway segments and trachealis smooth muscle strips studied in vitro, demonstrating that the effects of mechanical strain on airway reactivity reflect its direct effects on ASM<sup>45,48-52</sup>. Although the effects of deep inspiration on airway reactivity are short-lived, these observations suggest that mechanical strain could be а useful approach for suppressing hyperresponsiveness<sup>46,47,53,54</sup>.

We initially explored the effects of imposing mechanical strain on the airways for prolonged time periods to determine whether it could cause a longer term reduction of airway responsiveness. Chronic mechanical strain for 1-2 days applied to bronchial segments or tracheal muscle strips *in vitro* resulted in a decrease in their contractile responsiveness to ACh as assessed subsequently under unstrained conditions<sup>4</sup>. These results suggest that chronic strain can induce persistent alterations in the functional properties of the ASM tissues.

We subsequently tested the effects of chronic strain *in vivo* by applying CPAP to rabbits and ferrets for periods of 4 days to 2 weeks and found that CPAP suppressed airway reactivity to ACh *in* vivo<sup>1,2</sup>. Lobes,

airway segments and tracheal smooth muscle tissues excised from the lungs of these CPAP treated animals also exhibited reduced contractility *in vitro*. The effects of chronic mechanical strain on airway reactivity were persistent and could be detected for at least 24 hours after CPAP<sup>5</sup>. In addition, the continuous use of CPAP was not necessary for it to be effective: limiting CPAP to nocturnal periods for 4 days in rabbits was similarly effective in reducing airway responsiveness (Fig. 2A). We also tested the efficacy of chronic mechanical strain



at reducing airway hyperresponsiveness in the presence of allergic airway inflammation. In Ova-sensitized and challenged rabbits continuous CPAP administered for 4 days was effective at suppressing airway reactivity<sup>5</sup> (Fig 2B). We recently extended this study to human asthmatics: Adults with stable asthma and normal spirometry used nocturnal CPAP for 7 days<sup>6</sup>. CPAP resulted in a significant decrease in airway reactivity while a Sham-treated group of asthmatics had no significant change in airway reactivity.

# Effects of chronic mechanical strain on ASM phenotype and its responses to inflammatory mediators.

ASM cells in culture modulate their properties between a synthetic and differentiated phenotype<sup>84-86</sup>. Integrin proteins are widely recognized to be important regulators of cell phenotype, and can mediate transitions in the phenotypic status of cells in response to changes in the composition or stiffness of the extracellular matrix. Changes in ECM have been shown to modulate the secretion of eotaxin by ASM cells in

culture in response to stimulation with IL-13<sup>87</sup>.

Our data indicate that mechanical strain imposed on ASM tissues is a potent stimulus for regulating the phenotype and synthetic status ASM tissues<sup>14,15</sup>. When we imposed chronic mechanical strain on ASM tissues in vitro, the activation of pathways mediated by PI3-kinase dependent Akt were suppressed while the expression of smooth muscle phenotypespecific proteins was potentiated<sup>15</sup> (Fig. 4). We confirmed this effect on the airways of mice subjected to chronic mechanical strain in vivo: the activation of Akt was significantly depressed in animals subjected to prolonged high mechanical strain using PEEP as compared with controltreated animals (Fig. 13C)<sup>3</sup>. Because Akt is a critical mediator of pathways activated by inflammatory stimuli such as IL-13. we hypothesized that mechanical loads would suppress the inflammatory responses of ASM to local mediators and might thereby mitigate airway inflammation (Fig.4).



We performed studies on ASM tissues *in vitro* to evaluate the effects of mechanical strain on the responses of ASM tissues to stimulation with the inflammatory cytokine IL-13<sup>14,15</sup>. The administration of IL-13 to ASM tissues *in vitro* stimulated the synthesis and expression of the chemokine, eotaxin, and suppressed the expression of smooth muscle phenotype-specific proteins (Figs. 5,6). Subjecting ASM tissues to mechanical strain suppressed IL-13 stimulated eotaxin synthesis and secretion and potentiated the expression of smooth muscle specific proteins, promoting the differentiated phenotype. *Thus, while IL-13 promotes chemokine synthesis and the synthetic phenotype of ASM, mechanical strain opposes this effect, suppressing IL-13 stimulated eotaxin synthesis and promoting the differentiated phenotype. (Fig. 4)* 

Our studies have also established the role of integrin signaling in the regulation of ASM differentiation and mechano-sensitive signaling to the nucleus. We found that integrin-linked kinase (ILK), a multi-domain  $\beta$  integrin-binding protein kinase that regulates Akt, is a critical upstream regulator of signaling pathways that regulate the synthetic and differentiation functions of ASM tissues<sup>88</sup>. ILK forms a stable heterotrimeric complex with PINCH, an adaptor protein, and  $\alpha$ -parvin, which binds to actin filaments<sup>89</sup>. ILK also binds directly to  $\beta$  integrin proteins and to the mechano-sensitive adhesome protein paxillin, and paxillin binding is necessary for the localization of ILK to integrin adhesomes<sup>90</sup>. ILK regulates the PI3 kinase-dependent

activation of Akt<sup>91</sup>. We found that Akt activation inhibits the transcriptional regulator, serum response factor (srf) in ASM, thereby suppressing the expression of smooth muscle phenotypic proteins<sup>88</sup>. Mechanical loads inhibit the ILK- dependent activation of Akt, thus promoting the differentiated phenotype<sup>15</sup>(Fig. 4). Our preliminary data also show that the ILK complex also plays a critical role in regulating the mechanosensitivity of eotaxin synthesis in response to the stimulation of ASM with IL-13<sup>14</sup> (Fig. 10).

## Summary.

We have shown that chronic mechanical strain suppresses allergen-induced hyper-responsiveness *in vivo* in animal models of asthma and the effectiveness of nocturnal CPAP at reducing airway hyper-reactivity in adults with mild-moderate asthma. Our studies of ASM tissues indicate that mechanical strain is sensed and transduced by integrin adhesomes to signaling pathways that regulate the synthetic and differentiation status of ASM. Our proposed studies will use *in vitro* models to assess the effects of strain on the inflammatory responses of ASM tissues (*SA #1*), will evaluate the suppression of airway inflammation by chronic strain in murine models of asthma (*SA #2*), and will test the efficacy of mechanical strain as therapy to suppress airway inflammation and hyper-reactivity in children with severe asthma (*SA #3*).

# SPECIFIC AIM #3: DETERMINE WHETHER CPAP SUPPRESSES AIRWAY HYPER-REACTIVITY AND AIRWAY INFLAMMATION IN CHILDREN WITH SEVERE ASTHMA.

RATIONALE. Whereas some children with asthma have intermittent symptoms that are improved with short-acting bronchodilators, many have persistent symptoms requiring daily treatment with inhaled corticosteroids. Children with severe asthma often have ongoing symptoms, airway inflammation and hyperreactivity despite treatment with high doses of inhaled corticosteroids. They are at high risk for asthma exacerbation requiring systemic corticosteroids, emergency room visits and hospitalization. Children with severe asthma are often highly atopic with increased peripheral blood eosinophilia, aeroallergen sensitivity, elevated serum IgE concentrations, elevated eNO, and eosinophilia in induced sputum and BALF<sup>120-125</sup>. A novel non-pharmacologic treatment that suppresses airway hyper-reactivity and inflammation in children with severe asthma could provide a significant advance in the therapy for these difficult to treat patients. We hypothesize that chronic mechanical strain will suppress airway reactivity and inflammation in children with severe asthma. In SA #3 we will determine whether the use of nocturnal CPAP for 1 month in children with severe asthma suppresses airway reactivity as assessed by bronchial challenge, and airway inflammation by induced sputum.

PRELIMINARY DATA. Our recent study of adults with mild-moderate clinically stable asthma demonstrated that treatment with nocturnal CPAP for 1 week decreased airway reactivity (increase in  $PC_{20}$ ) compared to a Sham-treated group<sup>6</sup>. These results provided the pilot data for our current NIH phase II multi-center clinical trial designed to assess the effectiveness of using nocturnal CPAP to suppress airway reactivity in subjects with mild-moderate asthma. However, this trial is restricted primarily to adult patients who may not be steroid- dependent and are less likely to have persistent airway inflammation or exhibit airway remodeling. Therefore we plan to evaluate children with severe asthma, as CPAP therapy may be particularly beneficial to this group. Our study will also assess airway inflammation which is not included in previous or ongoing clinical trials.

# Fig.16. Nocturnal CPAP suppressed airway hyper-reactivity in an 8 yr old girl.

We assessed the effect of 1 month treatment with nocturnal CPAP (8 cm $H_2O$ ) or Sham (0 cm  $H_2O$ ) in two 8 year old girls who had  $PC_{20}$  <1 mg/ml, which is indicative of airway hyper-reactivity. The child treated with CPAP showed a marked decrease in airway reactivity (increased PC20), while the ham-treated child maintained airway. This demonstrates our ability to recruit and evaluate young children, and is consistent with our hypothesis.

#### 2.0 Inclusion/Exclusion Criteria

#### **SUBJECT RECRUITMENT**

#### **Inclusion Criteria:**

- 1. Children 8–17 yrs olds with severe asthma (N=120) will be recruited from the Pediatric High Risk Asthma Clinic and Pulmonary Clinics at Riley Hospital for Children at Indiana University Health.
- 2. Severe asthma will be defined by the need for medication therapies following steps 4-6 according to the National Institutes of Health's Asthma Care Quick Reference, September 2012 or high dose of inhaled corticosteroids.
- 3. Children on a stable regimen of asthma medications for at least 8 wks prior to enrollment without systemic corticosteroids for >4 wks will be eligible.

#### **Exclusion Criteria:**

- 1. Obese (>95% predicted BMI).
- 2. Congenital heart disease or chronic lung disease.
- 3. History of pneumothorax.
- 4. Inability to perform pulmonary function testing.
- 5. Oxygen saturation <93%.
- 6. FEV1 <70% predicted.
- 7. PC20 ≥16 mg/ml of methacholine.

#### 3.0 Enrollment/Randomization

# TREATMENT:

- 1. Nocturnal CPAP (8-12 cmH<sub>2</sub>O) or Sham (0 cmH<sub>2</sub>O).
- 2. Subjects will be randomized to use CPAP or Sham CPAP at night for a total of 28 days (+/- 3 days) with a minimum of 4 hrs/night for at least 5 days/wk. If patient is having asthma symptoms at time of final visit, treatment may be extended up to 14 additional days. If patient receives oral steroids at any time during treatment with nocturnal CPAP, the final visit will be extended to at least 21 days (3 weeks) after the last dose of oral steroid was given. Adherence to the use of CPAP will be checked by having the patient mail the SD data card from their machine to the Investigator on day 7 and day 14 of CPAP usage and by downloading the data at the time of the final visit. Adherence and tolerance of CPAP will be evaluated by periodic phone calls and documented daily calendar diary with hours of use.

# 4.0 Study Procedures:

- **1. Spirometry**: Spirometry will be performed after withholding bronchodilators. Forced vital capacity (FVC) and forced expiratory volume in 1 second ( $FEV_1$ ) will be measured using ATS guidelines.
- 2. Airway Reactivity assessed by MCh Bronchial Challenge: Testing will use the 5 breath dosimeter protocol recommended by ATS<sup>126</sup>. Following inhalation of saline, MCh will be inhaled in quadrupling concentrations starting with 0.0625 mg/ml and continuing until the MCh concentration required for FEV<sub>1</sub> to decrease by 20% from baseline (PC<sub>20</sub>) is achieved or a maximum MCh concentration of 16 mg/ml is inhaled.
- **3. Airway Inflammation assessed by Exhaled Nitric Oxide (eNO):** eNO will be measured at a constant expiratory flow of 50 ml/s with a chemiluminescence analyzer (NIOX; Aerocrine) using ATS quidelines<sup>127</sup>.
- **4. Airway Inflammation assessed by Induced Sputum**. Sputum induction will be performed after MCh challenge and treatment with albuterol to return FEV₁ to ≥ 70% predicted. Sputum will be induced by inhaling increasing concentrations (3 to 7%) of saline at 5 min intervals. Oscillating positive expiratory pressure (PEP) therapy may be used if needed to assist with sputum expectoration in conjunction with

saline treatments for up to 20 min or until an adequate sample is produced. Spirometry is performed after each expectoration to check that the  $FEV_1$  has not decreased by >20%, in which case the child would be given bronchodilator and no more hypertonic saline. Sputum will be processed for differential cell counts and supernatants stored at -80°C for subsequent analysis of eotaxin and eosinophil cationic protein<sup>128</sup>.

- **5. Asthma Symptom control:** Asthma control will be assessed by using the Asthma Control Test<sup>129</sup>.
- **6. Berlin score:** Questionnaire will be used to determine high or low risk status for obstructive sleep apnea<sup>130</sup>.

#### 5.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

#### **Adverse Events**

An adverse event (AE) is any untoward medical occurrence in a clinical investigation of a patient that does not necessarily have a causal relationship with the treatment. An AE is therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the administration of an investigational product, whether or not related to that investigational product.

The Investigator will probe, via discussion with the subject, for the occurrence of AEs during each subject visit and record the information in the site's source documents. Adverse events will be recorded in the subject internal data collection forms. Adverse events will be described by duration (start and stop dates and times), severity, outcome, treatment and relation to study medication, or if unrelated, the cause.

#### Serious Adverse Experiences (SAE)

An SAE is defined as any untoward medical occurrence that:

- Results in death
- Is considered life threatening (i.e., in the view of the investigator the adverse experience places the subject at immediate risk of death from the reaction, as it occurred; it does not include a reaction that, had it occurred in a more severe form, might have caused death)
- Requires hospital admission or prolongation of an existing hospitalization
- Results in persistent or significant disability/incapacity (i.e., a substantial disruption of a person's ability to conduct normal life functions)
- Is a congenital anomaly/birth defect
- Is an important medical event (i.e., when based upon appropriate medical judgment, the adverse experience may jeopardize the subject and may require medical or surgical intervention to prevent one of the above listed outcomes)

## **Data Safety Monitoring Plan**

Data Safety Monitor Gregory Montgomery, MD will monitor this study on an annual basis. Data to be monitored includes: data quality, subject recruitment, accrual and retention and adverse events. The results of related studies that impact subject safety and privacy will also be assessed.

Data monitoring will also include the interpretation of the data and confirming that the data is kept in a secure database. The co-investigators of the study will be doing an interim analysis and interpretation of the data on an annual basis.

Adverse events will be dealt with on a case by case basis and all institutions (IRB/ NIH) involved in the study will be notified by either a formal letter or memo.

The following information will be reported to the IRB on an annual basis with the continuing review:

- 1. Dates of monitoring
- 2. Summary of cumulative adverse events

- 3. Assessment of external factors that impact the safety of subjects
- 4. Summary of subject privacy and research data confidentiality
- 5. Any changes in risk-benefit ratio

## 6.0 Study Withdrawal/Discontinuation

If the parent/guardian chooses to withdraw the subject from the study, then the parent/guardian will inform a member of the research team. At that time, no further testing will be obtained. Samples already obtained from the subject prior to withdrawal will still be included in analysis.

**Management of Increased Asthma Symptoms**: If a subject's asthma symptoms worsen during the course of the treatment period, they will be directed to their pediatric pulmonologist or the High Risk Asthma clinic for management. Any changes in therapy, including controller medications or courses of systemic steroids will be recorded. As the enrolled subjects have severe asthma, one course of systemic steroids in 4 weeks would not be considered unusual and would not trigger withdrawal from the study. However, an inpatient hospitalization or two courses of systemic steroids in the 4 week treatment period will trigger withdrawal from the study

## 7.0 Statistical Considerations

#### ANALYSIS:

**Primary Outcome**: The change in airway reactivity (logPC20) measured prior to and after 4 wks of either CPAP or SHAM treatment. We will compare the change in PC20 between two groups using an analysis of covariance (ANCOVA) model, adjusting for baseline PC20. We anticipate that PC20 will increase for the CPAP treated group, but not change for the SHAM treated subjects.

**Secondary Outcomes**: Airway Inflammation assessed as the change in the percentage eosinophils in the induced sputum measured prior to and after 4 wks CPAP or SHAM treatment. We will compare the change between two groups using an ANCOVA model adjusting for baseline percentage eosinophils. We anticipate that eosinophilia will decrease for the CPAP treated group, but not in the SHAM treated subjects.

Justification of Sample Size: Change in Airway Responsiveness: We calculated the sample size based on the difference of logPC20 changes between groups. Our previous study showed a difference of change in logPC20 between CPAP and SHAM groups as 0.41 with a standard deviation of 0.46. With a 1 month intervention period in our study (compared to 1 week in previous study), we expect a larger effect size. Therefore, we conservatively assume a 0.41 difference and a 0.46 standard deviation. With 30 patients in each group, we expect 27 of them will complete the study. We will have more than 85% power to detect such a difference with a 5% Type I error rate using a two-sample t-test. ANCOVA model will be more powerful than the t-test. Change in Airway Inflammation: We calculated the smallest changes in airway inflammation that can be detected with the sample size generated above. With 27 patients completing the study, we have 80% power to detect an effect size as small as 78% (difference of changes is 78% of the standard deviation) using a t-test.

#### ANTICIPATED RESULTS.

Based upon our previous experience that CPAP suppresses airway reactivity in adults with mild-moderate asthma, our preliminary data in children and our animal models, we anticipate that nocturnal CPAP will suppress airway reactivity in children with severe asthma. These findings would have important clinical implications and justify a multi-center trial for much longer periods of CPAP treatment to evaluate its potential in decreasing asthma symptoms and medication usage in children with severe asthma.

We also expect CPAP to suppress airway inflammation. Although our primary measurement of airway inflammation is induced sputum eosinophilia, we will evaluate additional inflammatory markers. It is possible that our sample size will be too small to obtain statistical significance for these markers. However, if we find that CPAP shows a tendency to decrease airway inflammation, our results could be used to power a larger clinical trial. It is possible that CPAP will increase airway inflammation, but this seems unlikely as

CPAP in adults with obstructive sleep apnea has been found to decrease systemic inflammatory markers 131,132.

# 8.0 Privacy/Confidentiality Issues

Each study subject will be assigned a subject number. All samples will be identified only by subject number when submitted to the research laboratory for analysis. The enrollment list containing both the subject number and identifiable information will be kept on a password protected server.

### Security and confidentiality

To comply with HIPAA guidelines, processes and procedures have been documented and implemented to ensure the security and protection of the study data within the computer operations center, the server, and the database. IU uses a three level security model to secure and protect data collected and stored within REDCap. This model is as follows: 1) an individual must register an account within the Indiana CTSI Hub and either be assigned a username/password if external to IU or use their IU login credentials and authenticate via IU's Central Authentication Service (CAS); 2) once a Hub account has been established, an individual must submit a request for a REDCap account; the request must be approved and then a REDCap account is established; and, 3) an individual must have their REDCap account be granted appropriate access and privileges to the specific project database by the project PI or delegate. In addition, since REDCap is webbased, IU utilizes SSL (https) encryption for secure connectivity.

# 9.0 Follow-up and Record Retention

#### **Enrollment:**

Enrolling sufficient subjects is always challenging; however we were successful at this in our previous CPAP study<sup>6</sup>. Riley Hospital for Children is the primary referral center for all of Indiana and our pediatric pulmonary group manages most of the severe pediatric asthma, so we do not expect problems recruiting subjects for this study. In multiple previous studies we recruited more than 100 subjects <sup>133-137</sup>.

# **CPAP Measures:**

In our preliminary studies, the use of CPAP for an average of 4 hrs/night was effective. Our CPAP devices can monitor the number of hours that CPAP is actually being used by measuring respiratory pressure fluctuations. Daily usage statistics can be stored on an SD card that is downloaded after 1 week, 2 weeks and 4 weeks of treatment. To reinforce adherence, we insure mask comfort at the initial visit, use humidification to prevent nasal drying and reinforce adherence with regular telephone calls and documented daily calendar diary with of hours of use.

#### **Data Capture System**

The Research Electronic Data CAPture (REDCap) database system will be used to collect data for this study. The REDCap software toolset provides a secure, web-based environment that is flexible enough to be used for a variety of types of research, provides an intuitive interface for users to enter data and have real time validation rules (with automated data type and range checks) at the time of entry. The system offers easy data manipulation with logged auditing, functionality for reporting, monitoring and querying patient records, and an automated export mechanism to common statistical packages such as: SPSS, SAS, Stata, R/S-Plus. REDCap has been used within Indiana University and affiliates since April 2009 and it currently supports 177 projects and over 380 users within IU, Purdue, Notre Dame, IU Health, VA, Rehabilitation Hospital of Indiana, and Wishard Health. The input data will be stored in secured server for storage and analysis.

#### Backup

At all times, appropriate backup copies of the database and related software files will be maintained and the information will be appropriately protected from illegitimate access. At critical junctures of the protocol (e.g.,

production of interim reports and final reports), a permanent archive of the database will be made. Archived versions of the database will be saved for at least three years after the end of the study.

# Availability and Retention of Investigational Records:

The Investigator must make study data accessible to authorized representatives of the NIH and IRB/IEC upon request. A file for each subject must be maintained that includes the signed Informed Consent, HIPAA Authorization and copies of all source documentation related to that subject. The Investigator must ensure the reliability and availability of source documents from which the information on the internal data collection forms was derived. All study documents (subject files, signed informed consent forms, copies of internal data collection forms, Study File Notebook, etc.) must be kept secured for a period of three years.

## 10.0 ADMINISTRATIVE, ETHICAL, REGULATORY CONSIDERATIONS

The study will be conducted according to the Declaration of Helsinki, Protection of Human Volunteers (21 CFR 50), Institutional Review Boards (21 CFR 56), and Obligations of Clinical Investigators (21 CFR 312).

To maintain confidentiality, all lung function data, evaluation forms, reports and other records will be identified by a coded number and initials only. All study records will be kept in a locked file cabinet and code sheets linking a subject's name to a subject identification number will be stored separately in another locked file cabinet. Clinical information will not be released without written permission of the subject, except as necessary for monitoring by the FDA. The Investigator must also comply with all applicable privacy regulations (e.g., Health Insurance Portability and Accountability Act of 1996, EU Data Protection Directive 95/46/EC).

#### **Protocol Amendments**

Any amendment to the protocol will be written by the Study Principal Investigators and submitted to the IRB for their approval.

#### **Publications**

The preparation and submittal for publication of manuscripts containing the study results shall be in accordance with a process determined by mutual written agreement among the study Sponsor and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to, the Health Insurance Portability and Accountability Act of 1996.

#### LITERATURE CITED

- 1. Xue Z, Zhang L, Ramchandani R, Liu Y, Antony VB, Gunst SJ and Tepper RS. Respiratory system responsiveness in rabbits in vivo is reduced by prolonged continuous positive airway pressure. *J Appl Physiol* 99: 677-682, 2005.
- 2. Xue Z, Zhang L, Liu Y, Gunst SJ and Tepper RS. Chronic inflation of ferret lungs with CPAP reduces airway smooth muscle contractility in vivo and in vitro. *J Appl Physiol* 104: 610-615, 2008.
- 3. Xue Z, Zhang W, Desai LP, Gao H, Gunst SJ and Tepper RS. Increased mechanical strain imposed on murine lungs during ventilation in vivo depresses airway responsiveness and activation of protein kinase Akt. *J Appl Physiol* 114: 1506-1510, 2013.
- 4. Tepper RS, Ramchandani R, Argay E., Zhang L, Xue Z, Liu Y and Gunst SJ. Chronic strain alters passive and contractile properties of rabbit airways. *J Appl Physiol* 98: 1949-1954, 2005.
- 5. Xue Z, Yu Y, Gao H, Gunst SJ and Tepper RS. Chronic continuous positive airway pressure (CPAP) reduces airway reactivity in vivo in an allergen-induced rabbit model of asthma. *J Appl Physiol* 111:353-357, 2011.
- 6. Busk M, Busk N, Puntenney P, Hutchins J, Yu Z, Gunst SJ and Tepper RS. Use of continuous positive airway pressure reduces airway reactivity in adults with asthma. *Eur Respir J* 41: 317-322, 2013.
- 7. Hirst SJ, Hallsworth MP, Peng Q and Lee TH. Selective induction of eotaxin release by interleukin-13 or interleukin-4 in human airway smooth muscle cells is synergistic with interleukin-1beta and is mediated by the interleukin-4 receptor alpha-chain. *Am J Respir Crit Care Med* 165: 1161-1171, 2002.
- 8. Laporte JC, Moore PE, Baraldo S, Jouvin MH, Church TL, Schwartzman IN, Panettieri RA, Jr., Kinet JP and Shore SA. Direct effects of interleukin-13 on signaling pathways for physiological responses in cultured human airway smooth muscle cells. *American Journal of Respiratory & Critical Care Medicine* 164: 141-148, 2001.
- 9. Grunstein MM, Hakonarson H, Leiter J, Chen M, Whelan R, Grunstein JS and Chuang S. IL-13-dependent autocrine signaling mediates altered responsiveness of IgE-sensitized airway smooth muscle. [see comments.]. *American Journal of Physiology Lung Cellular & Molecular Physiology* 282: L520-L528, 2002.
- Weldon D. The effects of corticosteroids on bone growth and bone density. Ann Allergy Asthma Immunol 103: 3-11, 2009.
- Kelly HW, Sternberg AL, Lescher R, Fuhlbrigge AL, Williams P, Zeiger RS, Raissy HH, Van Natta ML, Tonascia J and Strunk RC. Effect of inhaled glucocorticoids in childhood on adult height. N Engl J Med 367: 904-912, 2012.
- 12. <a href="http://www.fda.gov/Drugs/DrugSafety/InformationbyDrugClass/ucm199565.htm">http://www.fda.gov/Drugs/DrugSafety/InformationbyDrugClass/ucm199565.htm</a>. 8-17-2010.
- 13. Doeing DC and Solway J. Airway smooth muscle in the pathophysiology and treatment of asthma. *J Appl Physiol* 114: 834-843, 2013.
- 14. Desai, L, Tepper R.S, and Gunst S.J. IL-13 Stimulated Eotaxin release and Smooth muscle myosin heavy chain (SmMHC) expression are Inversely Modulated by Mechanical Load in Airway Smooth Muscle (ASM) Tissues. Am J Respir Crit Care Med . 2012.
- 15. Desai LP, Wu Y, Tepper RS and Gunst SJ. Mechanical stimuli and IL-13 interact at integrin adhesion complexes to regulate expression of smooth muscle myosin heavy chain in airway smooth muscle tissue. *Am J Physiol Lung Cell Mol Physiol* 301: L275-L284, 2011.
- Gavett SH, O'Hearn DJ, Karp CL, Patel EA, Schofield BH, Finkelman FD and Wills-Karp M. Interleukin-4 receptor blockade prevents airway responses induced by antigen challenge in mice. *American Journal of Physiology* 272: t-61, 1997.

- 17. Wills-Karp M. Immunologic basis of antigen-induced airway hyperresponsiveness. *Annual Review of Immunology* 17: 255-281, 1999.
- 18. Wills-Karp M, Luyimbazi J, Xu X, Schofield B, Neben TY, Karp CL and Donaldson DD. Interleukin-13: central mediator of allergic asthma. *Science* 282: 2258-2261, 1998.
- 19. Wills-Karp M. Interleukin-13 in asthma pathogenesis. *Immunol Rev* 202: 175-190, 2004.
- 20. Wills-Karp M, Gavett SH, Schofield B and Finkelman F. Role of interleukin-4 in the development of allergic airway inflammation and airway hyperresponsiveness. *Advances in Experimental Medicine & Biology* 409: 343-347, 1996.
- 21. Grunig G, Warnock M, Wakil AE, Venkayya R, Brombacher F, Rennick DM, Sheppard D, Mohrs M, Donaldson DD, Locksley RM and Corry DB. Requirement for IL-13 independently of IL-4 in experimental asthma. *Science* 282: 2261-2263, 1998.
- 22. Kuperman DA, Huang X, Koth LL, Chang GH, Dolganov GM, Zhu Z, Elias JA, Sheppard D and Erle DJ. Direct effects of interleukin-13 on epithelial cells cause airway hyper-reactivity and mucus overproduction in asthma. *Nature Medicine* 8: 885-889, 2002.
- 23. Hashimoto S, Gon Y, Takeshita I, Maruoka S and Horie T. IL-4 and IL-13 induce myofibroblastic phenotype of human lung fibroblasts through c-Jun NH2-terminal kinase-dependent pathway. *Journal of Allergy & Clinical Immunology* 107: 1001-1008, 2001.
- 24. Venkayya R, Lam M, Willkom M, Grunig G, Corry DB and Erle DJ. The Th2 lymphocyte products IL-4 and IL-13 rapidly induce airway hyperresponsiveness through direct effects on resident airway cells. *American Journal of Respiratory Cell & Molecular Biology* 26: 202-208, 2002.
- 25. Hakonarson H and Grunstein MM. Autocrine regulation of airway smooth muscle responsiveness. *Respiratory Physiology & Neurobiology* 137: 263-276, 2003.
- 26. Moore PE, Church TL, Chism DD, Panettieri RA, Jr. and Shore SA. IL-13 and IL-4 cause eotaxin release in human airway smooth muscle cells: a role for ERK. *Am J Physiol Lung Cell Mol Physiol* 282: L847-L853, 2002.
- 27. Akiho H, Blennerhassett P, Deng Y and Collins SM. Role of IL-4, IL-13, and STAT6 in inflammation-induced hypercontractility of murine smooth muscle cells. *Am J Physiol Gastrointest Liver Physiol* 282: G226-G232, 2002.
- 28. Eum SY, Maghni K, Tolloczko B, Eidelman DH and Martin JG. IL-13 may mediate allergen-induced hyperresponsiveness independently of IL-5 or eotaxin by effects on airway smooth muscle. *Am J Physiol Lung Cell Mol Physiol* 288: L576-L584, 2005.
- 29. Renauld JC. New insights into the role of cytokines in asthma. *J Clin Pathol* 54: 577-589, 2001.
- 30. Riffo-Vasquez Y and Spina D. Role of cytokines and chemokines in bronchial hyperresponsiveness and airway inflammation. *Pharmacol Ther* 94: 185-211, 2002.
- 31. Rosenberg HF, Phipps S and Foster PS. Eosinophil trafficking in allergy and asthma. *J Allergy Clin Immunol* 119: 1303-1310, 2007.
- 32. Chiba Y, Nakazawa S, Todoroki M, Shinozaki K, Sakai H and Misawa M. Interleukin-13 augments bronchial smooth muscle contractility with an up-regulation of RhoA protein. *Am J Respir Cell Mol Biol* 40: 159-167, 2009.
- 33. Lee JH, Kaminski N, Dolganov G, Grunig G, Koth L, Solomon C, Erle DJ and Sheppard D. Interleukin13 induces dramatically different transcriptional programs in three human airway cell types. *Am J Respir Cell Mol Biol* 25: 474-485, 2001.

- 34. Nelms K, Keegan AD, Zamorano J, Ryan JJ and Paul WE. The IL-4 receptor: signaling mechanisms and biologic functions. *Annual Review of Immunology* 17: 701-738, 1999.
- 35. Jiang H, Harris MB and Rothman P. IL-4/IL-13 signaling beyond JAK/STAT. *J Allergy Clin Immunol* 105: 1063-1070, 2000.
- 36. Richter A, Puddicombe SM, Lordan JL, Bucchieri F, Wilson SJ, Djukanovic R, Dent G, Holgate ST and Davies DE. The contribution of interleukin (IL)-4 and IL-13 to the epithelial-mesenchymal trophic unit in asthma. *American Journal of Respiratory Cell & Molecular Biology* 25: 385-391, 2001.
- 37. Hakonarson H, Maskeri N, Carter C and Grunstein MM. Regulation of TH1- and TH2-type cytokine expression and action in atopic asthmatic sensitized airway smooth muscle. *Journal of Clinical Investigation* 103: 1077-1087, 1999.
- 38. Hallsworth MP, Moir LM, Lai D and Hirst SJ. Inhibitors of mitogen-activated protein kinases differentially regulate eosinophil-activating cytokine release from human airway smooth muscle. *American Journal of Respiratory & Critical Care Medicine* 164: 688-697, 2001.
- 39. Moynihan B, Tolloczko B, Michoud MC, Tamaoka M, Ferraro P and Martin JG. MAP kinases mediate interleukin-13 effects on calcium signaling in human airway smooth muscle cells. *Am J Physiol Lung Cell Mol Physiol* 295: L171-L177, 2008.
- 40. Peng Q, Matsuda T and Hirst SJ. Signaling Pathways Regulating Interleukin-13-stimulated Chemokine Release from Airway Smooth Muscle. *American Journal of Respiratory and Critical Care Medicine* 169: 596-603, 2004.
- 41. An SS, Bai TR, Bates JH, Black JL, Brown RH, Brusasco V, Chitano P, Deng L, Dowell M, Eidelman DH, Fabry B, Fairbank NJ, Ford LE, Fredberg JJ, Gerthoffer WT, Gilbert SH, Gosens R, Gunst SJ, Halayko AJ, Ingram RH, Irvin CG, James AL, Janssen LJ, King GG, Knight DA, Lauzon AM, Lakser OJ, Ludwig MS, Lutchen KR, Maksym GN, Martin JG, Mauad T, McParland BE, Mijailovich SM, Mitchell HW, Mitchell RW, Mitzner W, Murphy TM, Pare PD, Pellegrino R, Sanderson MJ, Schellenberg RR, Seow CY, Silveira PS, Smith PG, Solway J, Stephens NL, Sterk PJ, Stewart AG, Tang DD, Tepper RS, Tran T and Wang L. Airway smooth muscle dynamics: a common pathway of airway obstruction in asthma. *Eur Respir J* 29: 834-860, 2007.
- 42. Weist A, Williams T, Kisling J, Clem C and Tepper RS. Volume history and effect on airway reactivity in infants and adults. *J Appl Physiol* 93: 1069-1074, 2002.
- 43. Skloot G, Permutt S and Togias A. Airway hyperresponsiveness in asthma: a problem of limited smooth muscle relaxation with inspiration. *J Clin Invest* 96: 2393-2403, 1995.
- 44. Scichilone N, Kapsali T, Permutt S and Togias A. Deep inspiration-induced bronchoprotection is stronger than bronchodilation. *Am J Respir Crit Care Med* 162: 910-916, 2000.
- 45. Shen X, Gunst SJ and Tepper RS. Effect of tidal volume and frequency on airway responsiveness in mechanically ventilated rabbits. *J Appl Physiol* 83: 1202-1208, 1997.
- 46. King GG, Moore BJ, Seow CY and Pare PD. Time course of increased airway narrowing caused by inhibition of deep inspiration during methacholine challenge. *Am J Respir Crit Care Med* 160: 454-457, 1999.
- 47. Kapsali T, Permutt S, Laube B, Scichilone N and Togias A. Potent bronchoprotective effect of deep inspiration and its absence in asthma. *J Appl Physiol* 89: 711-720, 2000.
- 48. Gunst SJ and Lai-Fook SJ. Effect of inflation on trachealis muscle tone in canine tracheal segments in vitro. *J Appl Physiol :Respirat Environ Exercise Physiol* 54: 906-913, 1983.
- 49. Gunst SJ, Stropp JQ and Service J. Mechanical modulation of pressure-volume characteristics of contracted canine airways in vitro. *J Appl Physiol* 68: 2223-2229, 1990.

- 50. Fredberg JJ, Inouye D, Miller B, Nathan M, Jafari S, Raboudi SH, Butler JP and Shore SA. Airway smooth muscle, tidal stretches, and dynamically determined contractile states. *Am J Respir Crit Care Med* 156: 1752-1759, 1997.
- 51. Wang L, Pare PD and Seow CY. Effects of length oscillation on the subsequent force development in swine tracheal smooth muscle. *J Appl Physiol* 88: 2246-2250, 2000.
- 52. Wang L, Pare PD and Seow CY. Effect of chronic passive length change on airway smooth muscle length-tension relationship. *J Appl Physiol* 90: 734-740, 2001.
- 53. Malmberg P, Larsson K, Sundblad BM and Zhiping W. Importance of the time interval between FEV1 measurements in a methacholine provocation test. *European Respiratory Journal* 6: 680-686, 1993.
- 54. Takeda M, Ito W, Tanabe M, Ueki S, Kato H, Kihara J, Tanigai T, Chiba T, Yamaguchi K, Kayaba H, Imai Y, Okuyama K, Ohno I, Sasaki T and Chihara J. Allergic airway hyperresponsiveness, inflammation, and remodeling do not develop in phosphoinositide 3-kinase gamma-deficient mice. *J Allergy Clin Immunol* 123: 805-812, 2009.
- 55. Kamm KE and Stull JT. The function of myosin and myosin light chain kinase phosphorylation in smooth muscle. *Annual Review of Pharmacology & Toxicology* 25: 593-620, 1985.
- 56. Gunst SJ. Applicability of the sliding filament/crossbridge paradigm to smooth muscle. [Review] [255 refs]. *Reviews of Physiology Biochemistry & Pharmacology* 134: 7-61, 1999.
- 57. Zhang W and Gunst SJ. Interactions of airway smooth muscle cells with their tissue matrix: implications for contraction. *Proc Am Thorac Soc* 5: 32-39, 2008.
- 58. Gunst SJ and Zhang W. Actin cytoskeletal dynamics in smooth muscle: a new paradigm for the regulation of smooth muscle contraction. *Am J Physiol Cell Physiol* 295: C576-C587, 2008.
- 59. Zhang W, Wu Y, Du L, Tang DD and Gunst SJ. Activation of the Arp2/3 complex by N-WASp is required for actin polymerization and contraction in smooth muscle. *Am J Physiol Cell Physiol* 288: C1145-C1160, 2005.
- 60. Zhang W and Gunst SJ. Dynamics of Cytoskeletal and Contractile Protein Organization: An Emerging Paradigm for Airway Smooth Muscle Contraction. In: Airway Smooth Muscle Biology and Pharmacology, edited by Chung KF. Wiley Press, 2008.
- 61. Zhang W and Gunst SJ. Interactions of Airway Smooth Muscle Cells with Their Tissue Matrix: Implications for Contraction. *Proc Am Thorac Soc* 5: 32-39, 2008.
- 62. Gunst SJ, Tang DD and Opazo SA. Cytoskeletal remodeling of the airway smooth muscle cell: a mechanism for adaptation to mechanical forces in the lung. *Respir Physiol Neurobiol* 137: 151-168, 2003.
- 63. Tang DD and Gunst SJ. Roles of focal adhesion kinase and paxillin in the mechanosensitive regulation of myosin phosphorylation in smooth muscle. *J Appl Physiol* 91: 1452-1459, 2001.
- 64. Tang DD, Mehta D and Gunst SJ. Mechanosensitive tyrosine phosphorylation of paxillin and focal adhesion kinase in tracheal smooth muscle. *Am J Physiol* 276: C250-8, 1999.
- 65. Mehta D, Wu MF and Gunst SJ. Role of contractile protein activation in the length-dependent modulation of tracheal smooth muscle force. *Am J Physiol* 270: C243-52, 1996.
- 66. Tang DD, Turner CE and Gunst SJ. Expression of non-phosphorylatable paxillin mutants in canine tracheal smooth muscle inhibits tension development. *J Physiol* 553: 21-35, 2003.
- 67. Nikolopoulos SN and Turner CE. Molecular dissection of actopaxin-integrin-linked kinase-Paxillin interactions and their role in subcellular localization. *J Biol Chem* 277: 1568-1575, 2002.
- 68. Tang DD, Wu MF, Opazo Saez AM and Gunst SJ. The focal adhesion protein paxillin regulates contraction in canine tracheal smooth muscle. *J Physiol (Lond)* 542: 501-513, 2002.
- 69. Schaller MD. Paxillin: a focal adhesion-associated adaptor protein. Oncogene 20: 6459-6472, 2001.

- 70. Tang DD and Gunst SJ. Depletion of focal adhesion kinase by antisense depresses contractile activation of smooth muscle. *Am J Physiol Cell Physiol* 280: C874-C883, 2001.
- 71. Turner CE. Paxillin and focal adhesion signalling. *Nature Cell Biology* 2: E231-E236, 2000.
- 72. Turner CE. Paxillin interactions. *J Cell Sci* 113 Pt 23: 4139-4140, 2000.
- 73. Sawada Y and Sheetz MP. Force transduction by Triton cytoskeletons. *Journal of Cell Biology* 156: 609-615, 2002.
- 74. Ingber DE. Tensegrity: the architectural basis of cellular mechanotransduction. *Annu Rev Physiol* 59:575-599, 1997.
- 75. Ingber DE. The mechanochemical basis of cell and tissue regulation. *Mech Chem Biosyst* 1: 53-68,2004.
- 76. Katsumi A, Orr AW, Tzima E and Schwartz MA. Integrins in Mechanotransduction. *J Biol Chem* 279:12001-12004, 2004.
- 77. Wang N, Butler JP and Ingber DE. Mechanotransduction across the cell surface and through the cytoskeleton. *Science* 260: 1124-1127, 1993.
- 78. Opazo Saez A., Zhang W, Wu Y, Turner CE, Tang DD and Gunst SJ. Tension development during contractile stimulation of smooth muscle requires recruitment of paxillin and vinculin to the membrane. *Am J Physiol Cell Physiol* 286: C433-C447, 2004.
- 79. Huang Y, Zhang W and Gunst SJ. Activation of vinculin induced by cholinergic stimulation regulates contraction of tracheal smooth muscle tissue. *J Biol Chem* 286(5): 3630-3644, 2010.
- 80. Zhang W, Wu Y, Wu C and Gunst SJ. Integrin-linked kinase (ILK) regulates N-WASp-mediated actin polymerization and tension development in tracheal smooth muscle. *J Biol Chem* 282: 34568-34580, 2007.
- 81. Zhang W, Huang Y and Gunst SJ. The small GTPase RhoA regulates the contraction of smooth muscle tissues by catalyzing the assembly of cytoskeletal signaling complexes at membrane adhesion sites. *J Biol Chem* 287: 33996-34008, 2012.
- 82. Seow CY and Fredberg JJ. Emergence of airway smooth muscle functions related to structural malleability. *J Appl Physiol* 110: 1130-1135, 2011.
- 83. Pratusevich VR, Seow CY and Ford LE. Plasticity in canine airway smooth muscle. *J Gen Physiol* 105:73-94, 1995.
- Halayko AJ and Solway J. Plasticity in Skeletal, Cardiac, and Smooth Muscle: Invited Review: Molecular mechanisms of phenotypic plasticity in smooth muscle cells. *J Appl Physiol* 90: 358-368, 2001.
- 85. Halayko AJ and Solway J. Molecular mechanisms of phenotypic plasticity in smooth muscle cells. *J Appl Physiol* 90: 358-368, 2001.
- 86. Halayko AJ, Camoretti-Mercado B, Forsythe SM, Vieira JE, Mitchell RW, Wylam ME, Hershenson MB and Solway J. Divergent differentiation paths in airway smooth muscle culture: induction of functionally contractile myocytes. *Am J Physiol* 276: L197-L206, 1999.
- 87. Hirst SJ, Twort CH and Lee TH. Differential effects of extracellular matrix proteins on human airway smooth muscle cell proliferation and phenotype. *Am J Respir Cell Mol Biol* 23: 335-344, 2000.
- 88. Wu Y, Huang Y, Herring BP and Gunst SJ. Integrin-linked kinase regulates smooth muscle differentiation marker gene expression in airway tissue. *Am J Physiol Lung Cell Mol Physiol* 295: L988-L997, 2008.

- 89. Wu C. Integrin-linked kinase and PINCH: partners in regulation of cell-extracellular matrix interaction and signal transduction. *J Cell Sci* 112 ( Pt 24): 4485-4489, 1999.
- 90. Nikolopoulos SN and Turner CE. Integrin-linked kinase (ILK) binding to paxillin LD1 motif regulates ILK localization to focal adhesions. *J Biol Chem* 276: 23499-23505, 2001.
- 91. Persad S, Attwell S, Gray V, Mawji N, Deng JT, Leung D, Yan J, Sanghera J, Walsh MP and Dedhar S. Regulation of protein kinase B/Akt-serine 473 phosphorylation by integrin-linked kinase: critical roles for kinase activity and amino acids arginine 211 and serine 343. *J Biol Chem* 276: 27462-27469, 2001.
- 92. Liu S, Slepak M and Ginsberg MH. Binding of Paxillin to the alpha 9 Integrin Cytoplasmic Domain Inhibits Cell Spreading. *J Biol Chem* 276: 37086-37092, 2001.
- 93. Guan JL. Focal adhesion kinase in integrin signaling. *Matrix Biology* 16: 195-200, 1997.
- 94. Hanks SK and Polte TR. Signaling through focal adhesion kinase. *Bioessays* 19: 137-145, 1997.
- 95. Tang DD, Zhang W and Gunst SJ. The adapter protein CrkII regulates neuronal Wiskott-Aldrich syndrome protein, actin polymerization, and tension development during contractile stimulation of smooth muscle. *J Biol Chem* 280: 23380-23389, 2005.
- 96. Tang DD and Gunst SJ. The small GTPase Cdc42 regulates actin polymerization and tension development during contractile stimulation of smooth muscle. *J Biol Chem* 279: 51722-51728, 2004.
- 97. Zhang W, Du L and Gunst SJ. The effects of the small GTPase RhoA on the muscarinic contraction of airway smooth muscle result from its role in regulating actin polymerization. *Am J Physiol Cell Physiol* 299: C298-C306, 2010.
- 98. Gunst SJ and Stropp JQ. Pressure-volume and length-stress relationships in canine bronchi in vitro. *J Appl Physiol* 64: 2522-2531, 1988.
- 99. Zhang YJ, Chen K, Tu YZ, Velyvis A, Yang YW, Qin J and Wu CY. Assembly of the PINCH-ILK-CH-ILKBP complex precedes and is essential for localization of each component to cell-matrix adhesion sites. *J Cell Sci* 115: 4777-4786, 2002.
- 100. Hayasaka H, Simon K, Hershey ED, Masumoto KH and Parsons JT. FRNK, the autonomously expressed C-terminal region of focal adhesion kinase, is uniquely regulated in vascular smooth muscle: analysis of expression in transgenic mice. *J Cell Biochem* 95: 1248-1263, 2005.
- 101. Parsons JT. Focal adhesion kinase: the first ten years. *J Cell Sci* 116: 1409-1416, 2003.
- 102. Kim DY, Park JW, Jeoung D and Ro JY. Celastrol suppresses allergen-induced airway inflammation in a mouse allergic asthma model. *Eur J Pharmacol* 612: 98-105, 2009.
- 103. Hoover WC, Zhang W, Xue Z, Gao H, Chernoff J, Clapp DW, Gunst SJ and Tepper RS. Inhibition of p21 activated kinase (PAK) reduces airway responsiveness in vivo and in vitro in murine and human airways. *PLoS One* 7: e42601, 2012.
- 104. Leigh R, Ellis R, Wattie JN, Hirota JA, Matthaei KI, Foster PS, O'Byrne PM and Inman MD. Type 2 cytokines in the pathogenesis of sustained airway dysfunction and airway remodeling in mice. Am J Respir Crit Care Med 169: 860-867, 2004.
- 105. Yao W, Chang J, Sehra S, Travers JB, Chang CH, Tepper RS and Kaplan MH. Altered cytokine production by dendritic cells from infants with atopic dermatitis. *Clin Immunol* 137: 406-414, 2010.

- 106. Sehra S, Yao W, Nguyen ET, Ahyi AN, Tuana FM, Ahlfeld SK, Snider P, Tepper RS, Petrache I, Conway SJ and Kaplan MH. Periostin regulates goblet cell metaplasia in a model of allergic airway inflammation. *J Immunol* 186: 4959-4966, 2011.
- 107. Duguet A, Wang CG, Gomes R, Ghezzo H, Eidelman DH and Tepper RS. Greater velocity and magnitude of airway narrowing in immature than in mature rabbit lung explants. *Am J Respir Crit Care Med* 164: 1728-1733, 2001.
- 108. Tuck SA, Maghni K, Poirier A, Babu GJ, Periasamy M, Bates JH, Leguillette R and Lauzon AM. Time course of airway mechanics of the (+)insert myosin isoform knockout mouse. *Am J Respir Cell Mol Biol* 30: 326-332, 2004.
- 109. Andersson CK, Claesson HE, Rydell-Tormanen K, Swedmark S, Hallgren A and Erjefalt JS. Mice lacking 12/15-lipoxygenase have attenuated airway allergic inflammation and remodeling. *Am J Respir Cell Mol Biol* 39: 648-656, 2008.
- 110. Benayoun L, Letuve S, Druilhe A, Boczkowski J, Dombret MC, Mechighel P, Megret J, Leseche G, Aubier M and Pretolani M. Regulation of peroxisome proliferator-activated receptor gamma expression in human asthmatic airways: relationship with proliferation, apoptosis, and airway remodeling. *Am J Respir Crit Care Med* 164: 1487-1494, 2001.
- 111. Plant PJ, North ML, Ward A, Ward M, Khanna N, Correa J, Scott JA and Batt J. Hypertrophic airway smooth muscle mass correlates with increased airway responsiveness in a murine model of asthma. *Am J Respir Cell Mol Biol* 46: 532-540, 2012.
- 112. Rydell-Tormanen K, Uller L and Erjefalt JS. Remodeling of extra-bronchial lung vasculature following allergic airway inflammation. *Respir Res* 9: 18, 2008.
- 113. Zosky GR, von GC, Stumbles PA, Holt PG, Sly PD and Turner DJ. The pattern of methacholine responsiveness in mice is dependent on antigen challenge dose. *Respir Res* 5: 15, 2004.
- 114. Tomkinson A, Cieslewicz G, Duez C, Larson KA, Lee JJ and Gelfand EW. Temporal association between airway hyperresponsiveness and airway eosinophilia in ovalbumin-sensitized mice. *Am J Respir Crit Care Med* 163: 721-730, 2001.
- 115. Burchell JT, Wikstrom ME, Stumbles PA, Sly PD and Turner DJ. Attenuation of allergen-induced airway hyperresponsiveness is mediated by airway regulatory T cells. *Am J Physiol Lung Cell Mol Physiol* 296: L307-L319, 2009.
- 116. Branski RC, Perera P, Verdolini K, Rosen CA, Hebda PA and Agarwal S.
  Dynamic biomechanical strain inhibits IL-1beta-induced inflammation in vocal fold fibroblasts. J Voice 21: 651-660, 2007.
- 117. Smith KE, Metzler SA and Warnock JN. Cyclic strain inhibits acute pro-inflammatory gene expression in aortic valve interstitial cells. *Biomech Model Mechanobiol* 9: 117-125, 2010.
- 118. MacDonald KD, Chang HY and Mitzner W. An improved simple method of mouse lung intubation. *J Appl Physiol* 106: 984-987, 2009.
- 119. Brown RH, Walters DM, Greenberg RS and Mitzner W. A method of endotracheal intubation and pulmonary functional assessment for repeated studies in mice. *J Appl Physiol* 87: 2362-2365, 1999.
- 120. Fitzpatrick AM, Gaston BM, Erzurum SC and Teague WG. Features of severe asthma in schoolage children: Atopy and increased exhaled nitric oxide. *J Allergy Clin Immunol* 118: 1218-1225, 2006.
- 121. Fitzpatrick AM, Teague WG, Meyers DA, Peters SP, Li X, Li H, Wenzel SE, Aujla S, Castro M, Bacharier LB, Gaston BM, Bleecker ER and Moore WC. Heterogeneity of severe asthma in childhood: confirmation by cluster analysis of children in the National Institutes of Health/National Heart, Lung, and Blood Institute Severe Asthma Research Program. *J Allergy Clin Immunol* 127: 382-389, 2011.

- 122. Fitzpatrick AM, Baena-Cagnani CE and Bacharier LB. Severe asthma in childhood: recent advances in phenotyping and pathogenesis. *Curr Opin Allergy Clin Immunol* 12: 193-201, 2012.
- 123. Cowan K and Guilbert TW. Pediatric asthma phenotypes. *Curr Opin Pediatr* 24: 344-351, 2012.
- 124. Chipps BE, Szefler SJ, Simons FE, Haselkorn T, Mink DR, Deniz Y and Lee JH. Demographic and clinical characteristics of children and adolescents with severe or difficult-to-treat asthma. *J Allergy Clin Immunol* 119: 1156-1163, 2007.
- 125. Haselkorn T, Szefler SJ, Simons FE, Zeiger RS, Mink DR, Chipps BE, Borish L and Wong DA. Allergy, total serum immunoglobulin E, and airflow in children and adolescents in TENOR. *Pediatr Allergy Immunol* 21: 1157-1165, 2010.
- 126. Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE and Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. *Am J Respir Crit Care Med* 161: 309-329, 2000.
- 127. ATS Workshop Proceedings: Exhaled Nitric Oxide and Nitric Oxide Oxidative Metabolism in Exhaled Breath Condensate. Proceedings of the American Thoracic Society 3(2), 131-145. 2006.
- Lex C, Payne DN, Zacharasiewicz A, Li AM, Wilson NM, Hansel TT and Bush A. Sputum induction in children with difficult asthma: safety, feasibility, and inflammatory cell pattern. *Pediatr Pulmonol* 39: 318-324, 2005.
- 129. Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ and Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. *J Allergy Clin Immunol* 113: 59-65, 2004.
- 130. Netzer NC, Stoohs RA, Netzer CM, Clark K and Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. *Ann Intern Med* 131: 485-491, 1999.
- 131. Alonso-Fernandez A, Garcia-Rio F, Arias MA, Hernanz A, de la Pena M, Pierola J, Barcelo A, Lopez- Collazo E and Agusti A. Effects of CPAP on oxidative stress and nitrate efficiency in sleep apnoea: a randomised trial. *Thorax* 64: 581-586, 2009.
- 132. Arias MA, Garcia-Rio F, Alonso-Fernandez A, Hernanz A, Hidalgo R, Martinez-Mateo V, Bartolome S and Rodriguez-Padial L. CPAP decreases plasma levels of soluble tumour necrosis factor-alpha receptor 1 in obstructive sleep apnoea. *Eur Respir J* 32: 1009-1015, 2008.
- 133. Yao W, Barbe-Tuana FM, Llapur CJ, Jones MH, Tiller C, Kimmel R, Kisling J, Nguyen ET, Nguyen J, Yu Z, Kaplan MH and Tepper RS. Evaluation of airway reactivity and immune characteristics as risk factors for wheezing early in life. *J Allergy Clin Immunol* 126: 483-488, 201.
- 134. Tepper RS, Llapur CJ, Jones MH, Tiller C, Coates C, Kimmel R, Kisling J, Katz B, Ding Y and Swigonski N. Expired nitric oxide and airway reactivity in infants at risk for asthma 6. *J Allergy Clin Immunol* 122: 760-765, 2008.
- 135. Kim YJ, Hall GL, Christoph K, Tabbey R, Yu Z, Tepper RS and Eigen H. Pulmonary diffusing capacity in healthy Caucasian children. *Pediatr Pulmonol* 47: 469-475, 2012.
- 136. Jones M, Castile R, Davis S, Kisling J, Filbrun D, Flucke R, Goldstein A, Emsley C, Ambrosius W and Tepper RS. Forced expiratory flows and volumes in infants. Normative data and lung growth. *Am J Respir Crit Care Med* 161: 353-359, 2000.
- 137. Eigen H, Bieler H, Grant D, Christoph K, Terrill D, Heilman DK, Ambrosius WT and Tepper RS. Spirometric pulmonary function in healthy preschool children. *Am J Respir Crit Care Med* 163: 619-623, 2001.